CLINICAL TRIAL: NCT02340221
Title: A Phase III, Double-Blind, Placebo-Controlled, Randomized Study of Taselisib Plus Fulvestrant Versus Placebo Plus Fulvestrant in Postmenopausal Women With Estrogen Receptor-Positive and HER2-Negative Locally Advanced or Metastatic Breast Cancer Who Have Disease Recurrence or Progression During or After Aromatase Inhibitor Therapy
Brief Title: A Study of Taselisib + Fulvestrant Versus Placebo + Fulvestrant in Participants With Advanced or Metastatic Breast Cancer Who Have Disease Recurrence or Progression During or After Aromatase Inhibitor Therapy
Acronym: SANDPIPER
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The Sponsor discontinued the manufacturing and development of taselisib due to modest clinical benefit and limited tolerability.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GO29058; 2014-003185-25 (EudraCT Number)
Record Dates: First submitted 2015-01-13; First posted 2015-01-16 (Estimated); Results first posted 2019-01-25 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — 2-(3-(2-(1-isopropyl-3-methyl-1H-1,2-4-triazol-5-yl)-5,6-dihydrobenzo(f)imidazo(1,2-d)(1,4)oxazepin-9-yl)-1H-pyrazol-1-yl)-2-methylpropanamide; Fulvestrant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Taselisib + Fulvestrant (Experimental): Participants received taselisib 4 milligrams (mg) taken orally QD beginning at Cycle 1, Day 1 and fulvestrant 500 mg by IM injection at Cycle 1, Days 1 and 15, and then on Day 1 of each subsequent 28-day cycle until disease progression, unacceptable toxicity, or study termination by the Sponsor.
  Interventions: Drug: Taselisib; Drug: Fulvestrant
- Placebo + Fulvestrant (Placebo Comparator): Participants received placebo taken orally once daily (QD) beginning at Cycle 1, Day 1, and fulvestrant 500 mg administered by intramuscular (IM) injection at Cycle 1, Days 1 and 15, and then on Day 1 of each subsequent 28-day cycle until disease progression, unacceptable toxicity, or study termination by the Sponsor.
  Interventions: Drug: Placebo; Drug: Fulvestrant

INTERVENTIONS:
Drug: Taselisib — Taselisib 4 mg was administered as two tablets of 2 mg each as per the schedule specified in the respective arm.
  Other Names: GDC-0032, RO5537381
  Arms: Taselisib + Fulvestrant
Drug: Placebo — Placebo matching to taselisib was administered as per the schedule specified in the respective arm.
  Arms: Placebo + Fulvestrant
Drug: Fulvestrant — Fulvestrant 500 mg was administered as two IM injections of 250 mg each as per the schedule specified in the respective arms.
  Other Names: Faslodex

SUMMARY:
This international, multicenter, randomized, double-blinded, placebo-controlled study is designed to compare the efficacy and safety of taselisib + fulvestrant with that of placebo + fulvestrant in postmenopausal women with estrogen receptor (ER)-positive, human epidermal growth factor receptor-2 (HER2)-negative, oncogene that encodes for phosphatidylinositol-4,5-bisphosphate 3-kinase (PIK3CA)-mutant, unresectable, locally advanced or metastatic breast cancer after recurrence or progression during or after an aromatase inhibitor (AI) therapy. There will be a 2:1 randomization to the taselisib arm versus the placebo arm. Enrollment will be enriched for participants with PIK3CA mutant tumors via central testing. The anticipated duration of the study is approximately 3.5 years.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women with histologically or cytologically confirmed locally advanced or metastatic estrogen receptor (ER) positive breast cancer
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Participants for whom endocrine therapy (example [e.g.], fulvestrant) is recommended and treatment with cytotoxic chemotherapy is not indicated at time of entry into the study
* Radiologic/objective evidence of recurrence or progression to the most recent systemic therapy for breast cancer
* Radiologic/objective evidence of breast cancer recurrence or progression while on or within 12 months of the end of adjuvant treatment with an aromatase inhibitor (AI), or progression while on or within 1 month of the end of prior AI treatment for locally advanced or metastatic breast cancer
* Measurable disease via Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 (v1.1) or non-measurable, evaluable disease with at least one evaluable bone lesion via RECIST v1.1
* Consent to provide a formalin-fixed, paraffin-embedded (FFPE) tumor tissue block (preferred) or a minimum of 20 (25 preferred) freshly cut unstained tumor slides from the most recently collected, available tumor tissue for oncogene that encodes for phosphatidylinositol-4,5-bisphosphate 3-kinase (PIK3CA)-mutation testing
* A valid cobas PIK3CA mutation result by central testing is required
* Adequate hematologic and end-organ function within 28 days prior to treatment initiation

Exclusion Criteria:

* Human epidermal growth factor receptor 2 (HER2)-positive disease by local laboratory testing (immunohistochemistry 3 positive [IHC 3+] staining or in situ hybridization positive)
* Prior treatment with fulvestrant
* Prior treatment with a phosphatidylinositol 3-kinase (PI3K) inhibitor, mammalian target of rapamycin (mTOR) inhibitor (e.g. everolimus), or protein kinase B (AKT) inhibitor
* Prior anti-cancer therapy within 2 weeks prior to Day 1 of Cycle 1
* Prior radiation therapy within 2 weeks prior to Day 1 of Cycle 1
* All acute treatment-related toxicity must have resolved to Grade less than or equal to (</=) 1 or be deemed stable by the Investigator
* Prior treatment with greater than (>) 1 cytotoxic chemotherapy regimen for metastatic breast cancer
* Concurrent hormone replacement therapy
* Known untreated or active central nervous system (CNS) metastases
* Type 1 or Type 2 diabetes mellitus requiring anti-hyperglycemic medications
* History of inflammatory bowel disease or active bowel inflammation
* Clinically significant cardiac or pulmonary dysfunction
* Clinically significant history of liver disease, including cirrhosis, current alcohol abuse, or current known active infection with human immunodeficiency virus (HIV), hepatitis B or C virus

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 631 (Actual)
Dates: Start 2015-04-09 (Actual); Primary Completion 2021-06-29 (Actual); Study Completion 2021-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (157):
- United States (16):
  - Arizona Oncology, Tucson, Arizona
  - Arizona Oncology Associates, P.C., Tucson, Arizona
  - Georgia Cancer Specialists - Northside, Atlanta, Georgia
  - Northwest Georgia Oncology Centers, a Service of WellStar Cobb Hospital, Marietta, Georgia
  - Ingalls Hospital, Harvey, Illinois
  - Maryland Oncology Hematology, Rochville, Maryland
  - Dana Farber Can Ins, Boston, Massachusetts
  - Mercy Hospitals East Communities d/b/a Mercy Hospital St. Louis, St Louis, Missouri
  - MSKCC at Basking Ridge, Basking Ridge, New Jersey
  - John Theurer Cancer Ctr at Hackensack Univ Medical Ctr, Hackensack, New Jersey
  - Memorial Sloan-Kettering; Cancer Center, Commack, New York
  - Memorial Sloan Kettering Cancer Center; Memorial Sloan Kettering; at Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Oregon Health & Science University; Knight Cancer Institute, Community Hematology Oncology, Beaverton, Oregon
  - Pinnacle Health, Harrisburg, Pennsylvania
- Australia (7):
  - Liverpool Hospital; Cancer Therapy Centre, Liverpool, New South Wales
  - Macquarie University Hospital, Macquarie Park, New South Wales
  - Newcastle Mater Misericordiae Hospital; Oncology, Waratah, New South Wales
  - Mater Hospital; Oncology, Brisbane, Queensland
  - Austin Hospital; Medical Oncology, Heidelberg, Victoria
  - Sunshine Hospital; Oncology Research, St Albans, Victoria
  - St John of God Murdoch Hospital; Oncology West, Murdoch, Western Australia
- Austria (4):
  - Lkh-Univ. Klinikum Graz; Klinik Für Innere Medizin I, Graz
  - Tiroler Landeskrankenanstalten Ges.M.B.H.; Abt. Für Gynäkologie, Innsbruck
  - Ordensklinikum Linz Barmherzige Schwestern; Abt. fur Innere Medizin 1, Linz
  - Medizinische Universität Wien; Univ.Klinik für Innere Medizin I, Vienna
- Bosnia and Herzegovina (2):
  - University Clinical Center of the Republic of Srpska, Banja Luka
  - Clinic of Oncology, University Clinical Center Sarajevo, Sarajevo
- Bulgaria (4):
  - Complex Oncological Center - Plovdiv, EOOD, Plovdiv
  - MHAT Nadezhda, Sofia
  - SHATO - Sofia, Sofia
  - SHATOD Dr. Marko Antonov Markov-Varna, EOOD, Varna
- Canada (7):
  - Cross Cancer Institute, Edmonton, Alberta
  - British Columbia Cancer Agency (Bcca) - Vancouver Cancer Centre, Vancouver, British Columbia
  - Grand River Hospital, Kitchener, Ontario
  - The Ottawa Hospital Cancer Centre; Oncology, Ottawa, Ontario
  - Sunnybrook Health Science Centre, Toronto, Ontario
  - McGill University; Sir Mortimer B Davis Jewish General Hospital; Oncology, Montreal, Quebec
  - Hospital Du Saint-Sacrement, Québec, Quebec
- China (5):
  - the First Hospital of Jilin University, Changchun
  - Jilin Cancer Hospital, Changchun
  - Jiangsu Cancer Hospital, Nanjing
  - Fudan University Shanghai Cancer Center, Shanghai
  - Zhejiang Cancer Hospital, Zhejiang
- Colombia (2):
  - Clinica del Country, Bogotá
  - Oncomedica S.A., Montería
- Czechia (3):
  - University Hospital; Oncology and Radiotherapy, Hradec Králové
  - Fakultni nemocnice Olomouc; Onkologicka klinika, Olomouc
  - Vseobecna fakultni nemocnice v Praze, Prague
- Finland (2):
  - KYS Sadesairaala; Syopatautien poliklinikka, Kuopio
  - Turku Uni Central Hospital; Oncology Clinics, Turku
- France (10):
  - Centre Jean Perrin; Hopital De Semaine, Clermont-Ferrand
  - Centre Georges François Leclerc; Service Pharmacie, Bp 77980, Dijon
  - Hopital Prive Drome Ardeche; Chir 2A 2B, Guilherand-Granges
  - CHD Vendée, La Roche-sur-Yon
  - Hopital Dupuytren; Oncologie Medicale, Limoges
  - Institut régional du Cancer Montpellier, Montpellier
  - Institut Curie; Oncologie Medicale, Paris
  - Ch Lyon Sud; Onco Secteur Jules Courmont, Pierre-Bénite
  - Pole de Cancerologie Prive Strasbourgeois, Strasbourg
  - Centre Alexis Vautrin; Oncologie Medicale, Vandœuvre-lès-Nancy
- Germany (7):
  - Hochwaldkrankenhaus; Abt.Gynäkologie Geburtshilfe u.Senologie, Bad Nauheim
  - Praxisklinik Krebsheilkunde für Frauen / Brustzentrum (Dres. Kittel/Klare), Berlin
  - Onkologische Schwerpunktpraxis Kurfürstendamm, Berlin
  - Universitätsklinikum Essen; Zentrum Für Frauenheilkunde, Essen
  - Kooperatives Mammazentrum Hamburg Krankenhaus Jerusalem, Hamburg
  - Klinikum der Universität München; Frauenklinik - Onkologie II, München
  - Klinikum Mutterhaus der Borromäerinnen, Innere Medizin I, Trier
- Greece (6):
  - Alexandras General Hospital of Athens; Oncology Department, Athens
  - IASO General Hospital of Athens, Athens
  - Univ General Hosp Heraklion; Medical Oncology, Heraklion
  - University Hospital of Patras Medical Oncology, Pátrai
  - Euromedical General Clinic of Thessaloniki; Oncology Department, Thessaloniki
  - Papageorgiou General Hospital; Medical Oncology, Thessaloniki
- Italy (10):
  - Istituto Nazionale Tumori Irccs Fondazione g. PASCALE;U.O.C. Oncologia Medica Senologica, Napoli, Campania
  - ARCISPEDALE S. MARIA NUOVA - REGGIO EMILIA; Struttura Semplice Coordinamento Breast Unit Integrata, Reggio Emilia, Emilia-Romagna
  - A.O. Universitaria S. Maria Della Misericordia Di Udine; Oncologia, Udine, Friuli Venezia Giulia
  - IRCCS Istituto Nazionale Per La Ricerca Sul Cancro (IST); Oncologia Medica A, Genoa, Liguria
  - Istituto Europeo Di Oncologia, Milan, Lombardy
  - Centro Catanese Di Oncologia; Oncologia Medica, Catania, Sicily
  - Azienda Ospedaliero-Universitaria Careggi; SOD Radioterapia, Florence, Tuscany
  - Azienda USL 9 Grosseto; Dipartimento Politiche del Farmaco, Grosseto, Tuscany
  - Azienda usl 5 Di Pisa-Ospedale Di Pontedera;U.O. Oncologia, Pontedera, Tuscany
  - AZ. Usll12 Veneziana-Ospedale Dell'angelo;Oncologia Medica, Mestre, Veneto
- Mexico (5):
  - Iem-Fucam, D.F.
  - Instituto Nacional De Cancerologia; Oncology; Tumores Mamarios, Distrito Federal
  - Consultorio de Medicina Especializada; Dentro de Condominio San Francisco, Mexico City
  - Hospital San Jose Del Tec. de Monterrey; Oncology, Monterrey
  - Oaxaca Site Management Organization, Oaxaca City
- Netherlands (2):
  - Medisch Centrum Alkmaar, Alkmaar
  - Ziekenhuis Rijnstate, Arnhem
- Peru (4):
  - Instituto Nacional de Enfermedades Neoplasicas, Lima
  - Clinica Internacional, Sede San Borja; Unidad de Investigacion de Clínica Internacional, Lima
  - Oncocenter Peru S.A.C.; Oncosalud, Lima
  - Instituto Regional de Enfermedades Neoplasicas - IREN Norte, Trujillo
- Poland (10):
  - Bialostockie Centrum Onkologii; Oddzial Onkologii Klinicznej, Bialystok
  - Centrum Onkologii w Bydgoszczy; Oddzial Kliniczny Onkologii, Bydgoszcz
  - Uniwersyteckie Centrum Kliniczne, Klinika Onkologii i Radioterapii, Gdansk
  - Przychodnia Lekarska KOMED, Roman Karaszewski, Konin
  - Szpital Uniwersytecki w Krakowie, Oddział Kliniczny Kliniki Onkologii, Krakow
  - Woj.Wielospecjalistyczne Centrum Onkologii i Traumatologii; Oddz.Hematologii Pododz.Chemioterapii, Lodz
  - Centrum Onkologii Ziemi LUBELSKIEJ im. Sw Jana z Dukli, I oddz. Chemioterapii, Lublin
  - Zachodniopomorskie Centrum Onkologii, Osrodek Innowacyjnosci, Rozwoju i Badan Klinicznych, Szczecin
  - Centrum Onkologii - Instytut im. Marii Skłodowskiej-Curie Klinika Nowotworów Piersi i Chirurgii, Warsaw
  - Wojewodzki Szpital Specjalistyczny; Osrodek Badawczo-Rozwojowy, Oddzial Chemioterapii, Wroclaw
- Portugal (5):
  - Hospital Garcia de Orta; Servico de Oncologia Medica, Almada
  - IPO de Lisboa; Servico de Oncologia Medica, Lisbon
  - Hospital da Luz; Departamento de Oncologia Medica, Lisbon
  - Hospital de Santa Maria; Servico de Oncologia Medica, Lisbon
  - IPO do Porto; Servico de Oncologia Medica, Porto
- Romania (4):
  - Institut of Oncology Al. Trestioreanu Bucharest; Oncology Department, Bucharest
  - Prof. Dr. I. Chiricuta Institute of Oncology, Cluj-Napoca
  - Oncology Center Sf. Nectarie, Craiova
  - Euroclinic Center of Oncology SRL, Iași
- Russia (6):
  - Moscow City Oncology Hospital #62, Moscovskaya Oblast, Moscow Oblast
  - Regional Clinical Oncology Dispensary; Surgery Dept, Thoracic, Arkhangelsk
  - Ivanovo Regional Oncology Dispensary, Ivanovo
  - Clinical Oncology Dispensary of Ministry of Health of Tatarstan, Kazan'
  - State Inst. Of Healthcare Orenburg Regional Clinical Oncology Dis, Orenburg
  - S-Pb clinical scientific practical center of specialized kinds of medical care (oncological), Saint Petersburg
- Institute for Onc/Rad Serbia, Belgrade, Serbia
- South Korea (9):
  - Inje university Haeundae Paik Hospital, Busan
  - Chungbuk National University Hospital, Cheongju-si
  - National Cancer Center, Goyang-si
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Ulsan University Hosiptal, Ulsan
- Spain (11):
  - Complejo Hospitalario Universitario de Santiago (CHUS) ; Servicio de Oncologia, Santiago de Compostela, LA Coruña
  - Hospital Universitario Puerta de Hierro; Servicio de Oncologia, Majadahonda, Madrid
  - Hospital Universitario de Canarias;servicio de Oncologia, San Cristóbal de La Laguna, Tenerife
  - Hospital de Cruces; Servicio de Oncologia, Bilbao, Vizcaya
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clínic i Provincial; Servicio de Hematología y Oncología, Barcelona
  - Centro Oncologico MD Anderson Internacional; Servicio de Oncologia, Madrid
  - Hospital Ramon y Cajal; Servicio de Oncologia, Madrid
  - HOSPITAL DE MADRID NORTE SANCHINARRO- CENTRO INTEGRAL ONCOLOGICO CLARA CAMPAL; Servicio de Oncologia, Madrid
  - Fundación IVO, Valencia
  - Hospital Universitario Miguel Servet; Servicio Oncologia, Zaragoza
- Sweden (3):
  - Uni Hospital Linkoeping; Dept. of Oncology, Linköping
  - Sodersjukhuset; Onkologkliniken, Stockholm
  - Akademiska sjukhuset, Onkologkliniken, Uppsala
- Taiwan (4):
  - VETERANS GENERAL HOSPITAL; Department of General Surgery, Taipei
  - National Taiwan Uni Hospital; General Surgery, Taipei
  - Mackay Memorial Hospital; Dept of Surgery, Taipei
  - Koo Foundation Sun Yat-Sen Cancer Center; Hemato-Oncology, Taipei
- Thailand (3):
  - Department of Surgery, King Chulalongkorn Memorial Hospital, Bangkok
  - Ramathibodi Hospital; Dept of Med.-Div. of Med. Onc, Bangkok
  - Maharaj Nakorn Chiang Mai Hospital; Department of Surgery/Head Neck and Breast Unit; Clinical Trial, Chiang Mai
- Turkey (Türkiye) (5):
  - Baskent University Adana Dr. Turgut Noyan Practice and Research Hospital; Medical Oncology, Adana
  - Trakya University Medical Faculty Research And Practice Hospital Medical Oncology Department, Edirne
  - Istanbul Uni Cerrahpasa Medical Faculty Hospital; Medical Oncology, Istanbul
  - Ege Uni Medical Faculty; Oncology Dept, Izmir
  - Hacettepe Uni Medical Faculty Hospital; Oncology Dept, Sihhiye/Ankara

REFERENCES:
- [Derived] Moein A, Jin JY, Wright MR, Wong H. Quantitative characterization of the effects of fulvestrant alone or in combination with taselisib (PI3Kinase inhibitor) on longitudinal tumor growth in patients with estrogen receptor-positive, HER2-negative, PIK3CA-mutant, advanced or metastatic breast cancer. Cancer Chemother Pharmacol. 2024 Sep;94(3):421-436. doi: 10.1007/s00280-024-04690-4. Epub 2024 Jun 27. PMID 38937298
- [Derived] Dent S, Cortes J, Im YH, Dieras V, Harbeck N, Krop IE, Wilson TR, Cui N, Schimmoller F, Hsu JY, He J, De Laurentiis M, Sousa S, Drullinsky P, Jacot W. Phase III randomized study of taselisib or placebo with fulvestrant in estrogen receptor-positive, PIK3CA-mutant, HER2-negative, advanced breast cancer: the SANDPIPER trial. Ann Oncol. 2021 Feb;32(2):197-207. doi: 10.1016/j.annonc.2020.10.596. Epub 2020 Nov 10. PMID 33186740

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 155 centers in 28 countries.
Pre-assignment Details: The study enrolled postmenopausal women with estrogen receptor-positive and human epidermal receptor 2 (HER2)-negative locally advanced or metastatic breast cancer who had disease recurrence or progression during or after aromatase inhibitor therapy. Randomization was stratified by three factors: 1) visceral versus non-visceral disease, 2) sensitivity versus non-sensitivity to most recent endocrine therapy, and 3) geographical region.
Groups:
- Placebo+Fulvestrant: Participants received placebo taken orally QD beginning at Cycle 1, Day 1, and fulvestrant 500 mg administered by IM injection at Cycle 1, Days 1 and 15, and then on Day 1 of each subsequent 28-day cycle until disease progression, unacceptable toxicity, or study termination by the Sponsor.
- Taselisib+Fulvestrant: Participants received taselisib 4 mg taken orally QD beginning at Cycle 1, Day 1 and fulvestrant 500 mg by IM injection at Cycle 1, Days 1 and 15, and then on Day 1 of each subsequent 28-day cycle until disease progression, unacceptable toxicity, or study termination by the Sponsor.
Period: Overall Study
Arm/Group | Placebo+Fulvestrant | Taselisib+Fulvestrant
Started | 214 | 417
Completed | 0 | 0
Not Completed | 214 | 417
Not completed — Death | 100 | 197
Not completed — Withdrawal by Participant | 24 | 37
Not completed — Lost to Follow-up | 4 | 15
Not completed — Reason Not Specified | 85 | 165
Not completed — Study Terminated by Sponsor | 1 | 3

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) population included all randomized participants regardless of whether they received any amount of study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo+Fulvestrant | Taselisib+Fulvestrant | Total
Number analyzed (Participants) | 214 | 417 | 631
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.7 (10.0) | 60.1 (9.9) | 60.3 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 214 | 417 | 631
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic or Latino | 166 | 334 | 500
  Hispanic or Latino | 26 | 48 | 74
  Not Stated | 15 | 15 | 30
  Unknown | 7 | 20 | 27
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 147 | 285 | 432
  Asian | 38 | 72 | 110
  Unknown | 14 | 30 | 44
  American Indian or Alaska Native | 13 | 24 | 37
  Black or African American | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 3 | 3
  Multiple | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS) as Assessed by Investigator Using Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 (v1.1) at Primary Analysis
Description: PFS was defined as the time from randomization to disease progression as determined by the investigator with the use of RECIST v1.1 or death due to any cause, whichever occurred earlier. Disease progression was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study, including baseline. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 millimeters (mm). For non-target lesions, disease progression was defined as unequivocal progression of existing lesions. The appearance of one or more new lesions was also considered progression.
Time Frame: From randomization until the first occurrence of disease progression or death from any cause, whichever occurs earlier (up to the 15 Oct 2017 data cutoff, approximately 2.5 years)
Population: Randomized participants with PIK3CA-mutant tumors, regardless of whether they received any amount of study treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo+Fulvestrant | Taselisib+Fulvestrant
Number analyzed (Participants) | 176 | 340
months | 5.39 [3.68 to 7.29] | 7.43 [7.26 to 9.07]
Statistical Analysis 1: Comparison: Placebo+Fulvestrant vs Taselisib+Fulvestrant; Test type: Superiority; p = 0.0037, Log Rank; Hazard Ratio (HR) = 0.70, 95% CI 2-sided [0.56 to 0.89]

2. Primary Outcome: PFS as Assessed by Investigator Using RECIST v1.1 at Final Analysis
Description: PFS was defined as the time from randomization to disease progression as determined by the investigator with the use of RECIST v1.1 or death due to any cause, whichever occurred earlier. Disease progression was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study, including baseline. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. For non-target lesions, disease progression was defined as unequivocal progression of existing lesions. The appearance of one or more new lesions was also considered progression.
Time Frame: From randomization until the first occurrence of disease progression or death from any cause, whichever occurs earlier (up to approximately 6.2 years)
Population: Randomized participants with PIK3CA-mutant tumors, regardless of whether they received any amount of study treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo+Fulvestrant | Taselisib+Fulvestrant
Number analyzed (Participants) | 176 | 340
months | 5.55 [3.75 to 7.33] | 8.05 [7.33 to 9.10]
Statistical Analysis 1: Comparison: Placebo+Fulvestrant vs Taselisib+Fulvestrant; Test type: Superiority; p = 0.0008, Log Rank; Hazard Ratio (HR) = 0.71, 95% CI 2-sided [0.58 to 0.87]

3. Secondary Outcome: Percentage of Participants With Objective Response (Partial Response [PR] Plus Complete Response [CR]), as Assessed Using RECIST v.1.1 at Primary Analysis
Description: PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters. CR was defined as disappearance of all target and non-target lesions and normalization of tumor marker levels (as applicable to non-target lesions).
Time Frame: as for outcome 1
Population: Randomized participants with PIK3CA-mutant tumors and measurable disease at baseline, regardless of whether they received any amount of study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo+Fulvestrant | Taselisib+Fulvestrant
Number analyzed (Participants) | 134 | 264
percentage of participants | 11.9 [7.1 to 18.3] | 28.0 [22.7 to 33.8]
Statistical Analysis 1: Comparison: Placebo+Fulvestrant vs Taselisib+Fulvestrant; Test type: Superiority; p = 0.0002, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 3.0, 95% CI 2-sided [1.6 to 5.4]

4. Secondary Outcome: Percentage of Participants With Objective Response (PR Plus CR), as Assessed Using RECIST v.1.1 at Final Analysis
Description: as for outcome 3
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo+Fulvestrant | Taselisib+Fulvestrant
Number analyzed (Participants) | 134 | 264
percentage of participants | 13.4 [8.2 to 20.2] | 31.1 [25.5 to 36.8]
Statistical Analysis 1: Comparison: Placebo+Fulvestrant vs Taselisib+Fulvestrant; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 3.1, 95% CI 2-sided [1.7 to 5.4]

5. Secondary Outcome: Overall Survival (OS) at Primary Analysis
Description: OS was defined as the time from the date of randomization to the date of death due to any cause.
Time Frame: From randomization up to death from any cause (up to the 15 Oct 2017 data cutoff, approximately 2.5 years)
Population: Randomized participants with PIK3CA-mutant tumors, regardless of whether they received any amount of study treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo+Fulvestrant | Taselisib+Fulvestrant
Number analyzed (Participants) | 176 | 340
months | 23.56 [18.00 to NA] — Upper limit of confidence interval was not estimable due to the low number of participants with events. | 26.81 [21.29 to NA] — Upper limit of confidence interval was not estimable due to the low number of participants with events.
Statistical Analysis 1: Comparison: Placebo+Fulvestrant vs Taselisib+Fulvestrant; Test type: Superiority; p = 0.4151, Log Rank; Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.58 to 1.25]

6. Secondary Outcome: OS at Final Analysis
Description: OS was defined as the time from the date of randomization to the date of death due to any cause.
Time Frame: From randomization up to death from any cause (up to approximately 6.2 years)
Population: Randomized participants with PIK3CA-mutant tumors, regardless of whether they received any amount of study treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo+Fulvestrant | Taselisib+Fulvestrant
Number analyzed (Participants) | 176 | 340
months | 27.93 [24.38 to NA] — Upper limit of confidence interval was not estimable due to the low number of participants with events. | 27.79 [24.25 to 33.35]
Statistical Analysis 1: Comparison: Placebo+Fulvestrant vs Taselisib+Fulvestrant; Test type: Superiority; p = 0.9974, Log Rank; Hazard Ratio (HR) = 1.00, 95% CI 2-sided [0.75 to 1.33]

7. Secondary Outcome: Percentage of Participants With Clinical Benefit, as Assessed According to RECIST v1.1 at Primary Analysis
Description: Clinical benefit was defined as objective response (PR+CR), or no disease progression lasting for more than or equal to (>/=) 24 weeks since randomization. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters. CR was defined as disappearance of all target and non-target lesions and normalization of tumor marker levels (as applicable to non-target lesions). Disease progression was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study, including baseline. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. For non-target lesions, disease progression was defined as unequivocal progression of existing lesions. The appearance of one or more new lesions was also considered progression.
Time Frame: as for outcome 1
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo+Fulvestrant | Taselisib+Fulvestrant
Number analyzed (Participants) | 134 | 264
percentage of participants | 37.3 [29.1 to 45.7] | 51.5 [45.3 to 57.7]
Statistical Analysis 1: Comparison: Placebo+Fulvestrant vs Taselisib+Fulvestrant; Test type: Superiority; Odds Ratio (OR) = 1.9, 95% CI 2-sided [1.2 to 2.9]

8. Secondary Outcome: Percentage of Participants With Clinical Benefit, as Assessed According to RECIST v1.1 at Final Analysis
Description: as for outcome 7
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo+Fulvestrant | Taselisib+Fulvestrant
Number analyzed (Participants) | 134 | 264
percentage of participants | 45.5 [37.2 to 54.3] | 59.5 [53.6 to 65.4]
Statistical Analysis 1: Comparison: Placebo+Fulvestrant vs Taselisib+Fulvestrant; Test type: Superiority; Odds Ratio (OR) = 1.9, 95% CI 2-sided [1.2 to 3.0]

9. Secondary Outcome: Duration of Objective Response, as Assessed by Investigator Using RECIST v1.1 at Primary Analysis
Description: Duration of objective response: the time from the first tumor assessment that supported the participant's objective response (CR or PR, whichever was first recorded) to first documented disease progression or death due to any cause, whichever occurred first. CR was defined as disappearance of all target and non-target lesions and normalization of tumor marker levels (as applicable to non-target lesions). PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters. Disease progression: at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study, including baseline. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. For non-target lesions, disease progression was defined as unequivocal progression of existing lesions. The appearance of one or more new lesions was also considered progression.
Time Frame: Time from the first occurrence of a documented objective response to the time of the first documented disease progression or death from any cause, whichever occurs earlier (up to the 15 Oct 2017 data cutoff, approximately 2.5 years)
Population: Randomized participants with PIK3CA-mutant tumors and measurable disease at baseline, regardless of whether they received any amount of study treatment. Data are reported for participants with responses.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo+Fulvestrant | Taselisib+Fulvestrant
Number analyzed (Participants) | 16 | 74
months | 7.23 [6.51 to NA] — Upper limit of confidence interval was not estimable due to the low number of participants with events. | 8.74 [5.72 to 11.24]
Statistical Analysis 1: Comparison: Placebo+Fulvestrant vs Taselisib+Fulvestrant; Test type: Superiority; p = 0.6708, Log Rank; Hazard Ratio (HR) = 0.77, 95% CI 2-sided [0.23 to 2.59]

10. Secondary Outcome: Duration of Objective Response, as Assessed by Investigator Using RECIST v1.1 at Final Analysis
Description: as for outcome 9
Time Frame: Time from the first occurrence of a documented objective response to the time of the first documented disease progression or death from any cause, whichever occurs earlier (up to approximately 6.2 years)
Population: as for outcome 9
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo+Fulvestrant | Taselisib+Fulvestrant
Number analyzed (Participants) | 18 | 82
months | 7.39 [4.67 to 23.95] | 8.97 [7.36 to 12.91]
Statistical Analysis 1: Comparison: Placebo+Fulvestrant vs Taselisib+Fulvestrant; Test type: Superiority; p = 0.8286, Log Rank; Hazard Ratio (HR) = 1.09, 95% CI 2-sided [0.51 to 2.35]

11. Secondary Outcome: PFS as Assessed by Blinded Independent Central Review (BICR) Using RECIST v1.1 at Primary Analysis
Description: PFS was defined as the time from randomization to disease progression as determined by BICR with the use of RECIST v1.1 or death due to any cause, whichever occurred earlier. Disease progression was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study, including baseline. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. For non-target lesions, disease progression was defined as unequivocal progression of existing lesions. The appearance of one or more new lesions was also considered progression.
Time Frame: as for outcome 1
Population: Randomized participants with PIK3CA-mutant tumors, regardless of whether they received any amount of study treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo+Fulvestrant | Taselisib+Fulvestrant
Number analyzed (Participants) | 176 | 340
months | 5.39 [3.68 to 9.23] | 8.97 [7.39 to 9.49]
Statistical Analysis 1: Comparison: Placebo+Fulvestrant vs Taselisib+Fulvestrant; Test type: Superiority; p = 0.0023, Log Rank; Hazard Ratio (HR) = 0.66, 95% CI 2-sided [0.51 to 0.86]

12. Secondary Outcome: PFS as Assessed by BICR Using RECIST v1.1 at Final Analysis
Description: as for outcome 11
Time Frame: as for outcome 2
Population: Randomized participants with PIK3CA-mutant tumors, regardless of whether they received any amount of study treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo+Fulvestrant | Taselisib+Fulvestrant
Number analyzed (Participants) | 176 | 340
months | 5.55 [3.68 to 9.30] | 9.20 [8.15 to 10.87]
Statistical Analysis 1: Comparison: Placebo+Fulvestrant vs Taselisib+Fulvestrant; Test type: Superiority; p = 0.0095, Log Rank; Hazard Ratio (HR) = 0.72, 95% CI 2-sided [0.56 to 0.92]

13. Secondary Outcome: Percentage of Participants With Adverse Events at Primary Analysis
Description: An adverse event was any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product, regardless of causal attribution.
Time Frame: From randomization up to the 15 Oct 2017 data cutoff, approximately 2.5 years.
Population: The safety-evaluable population included all randomized participants who received at least one dose of taselisib or placebo or fulvestrant.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo+Fulvestrant | Taselisib+Fulvestrant
Number analyzed (Participants) | 213 | 416
percentage of participants | 89.7 | 95.4

14. Secondary Outcome: Percentage of Participants With Adverse Events at Final Analysis
Description: as for outcome 13
Time Frame: From randomization up to approximately 6.2 years
Population: as for outcome 13
Measure: Number; unit: percentage of participants
Arm/Group | Placebo+Fulvestrant | Taselisib+Fulvestrant
Number analyzed (Participants) | 213 | 416
percentage of participants | 91.1 | 97.1

15. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Taselisib
Time Frame: 1 to 4 hours (hrs) post-dose on Cycle (C) 1, Day (D) 1; 0 to 3 hrs pre-dose and 2 to 6 hrs post dose on Cycle 2, Day 1 (each cycle=28 days)
Population: The Pharmacokinetic (PK) population included all participants who received at least one dose of taselisib and provided valid (adequately documented dose time and PK sample time) PK assessments.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Taselisib+Fulvestrant
Number analyzed (Participants) | 417
ng/mL
  C1D1 | 18.2 (14.6)
  C2D1: number analyzed (Participants) | 359
  C2D1 | 66.6 (35.2)

16. Secondary Outcome: Minimum Observed Plasma Concentration (Cmin) of Taselisib
Time Frame: 1 to 4 hrs post-dose on Cycle 1, Day 1; 0 to 3 hrs pre-dose and 2 to 6 hrs post dose on Cycle 2, Day 1; 0 to 3 hrs pre-dose on Cycle 6, Day 1 (each cycle=28 days)
Population: The PK population included all participants who received at least one dose of taselisib and provided valid (adequately documented dose time and PK sample time) PK assessments.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Taselisib+Fulvestrant
Number analyzed (Participants) | 417
ng/mL
  C2D1: number analyzed (Participants) | 377
  C2D1 | 42.8 (26.6)
  C6D1: number analyzed (Participants) | 213
  C6D1 | 35.3 (31.5)

17. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire Core 30 (QLQ-C30) Score
Description: The EORTC QLQ-C30 consists of 30 questions that comprise aspects of participant's functioning assessment (physical, emotional, role, cognitive, and social); symptom scales (fatigue; nausea, vomiting, and pain; the global health/quality of life [QoL]); and single items (dyspnoea, insomnia, appetite loss, constipation, diarrhoea, and financial difficulties), within a recall period of "the past week." Most questions used a 4-point scale (1=Not at all to 4=Very much; two questions used a 7-point scale (1=Very poor to 7=Excellent). Scores were averaged and transformed to a 0-100 scale; a higher score for Global Qol/functional scales=better level of functioning; a higher score for symptom scale=greater degree of symptoms.
Time Frame: Baseline, C2D1 up to C7D1 (each cycle=28 days)
Population: Randomized participants with PIK3CA-mutant tumors, regardless of whether they received any amount of study treatment. Data are reported for evaluable participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo+Fulvestrant | Taselisib+Fulvestrant
Number analyzed (Participants) | 176 | 340
score on a scale
  Appetite Loss: Baseline: number analyzed (Participants) | 159 | 312
  Appetite Loss: Baseline | 15.9 (25.9) | 15.3 (23.3)
  Appetite Loss: Change at C2D1: number analyzed (Participants) | 147 | 292
  Appetite Loss: Change at C2D1 | -0.2 (25.7) | 6.2 (26.2)
  Appetite Loss: Change at C3D1: number analyzed (Participants) | 117 | 260
  Appetite Loss: Change at C3D1 | -4.3 (27.2) | 8.7 (28.1)
  Appetite Loss: Change at C4D1: number analyzed (Participants) | 100 | 231
  Appetite Loss: Change at C4D1 | -1.7 (26.1) | 8.4 (28.1)
  Appetite Loss: Change at C5D1: number analyzed (Participants) | 75 | 206
  Appetite Loss: Change at C5D1 | -0.4 (26.6) | 6.0 (27.2)
  Appetite Loss: Change at C6D1: number analyzed (Participants) | 66 | 171
  Appetite Loss: Change at C6D1 | -0.5 (22.3) | 6.6 (27.2)
  Appetite Loss: Change at C7D1: number analyzed (Participants) | 58 | 145
  Appetite Loss: Change at C7D1 | -5.7 (28.7) | 4.6 (26.5)
  Cognitive Functioning: Baseline: number analyzed (Participants) | 160 | 312
  Cognitive Functioning: Baseline | 85.3 (18.1) | 85.9 (18.7)
  Cognitive Functioning: Change at C2D1: number analyzed (Participants) | 147 | 292
  Cognitive Functioning: Change at C2D1 | 0.7 (16.5) | -1.1 (16.8)
  Cognitive Functioning: Change at C3D1: number analyzed (Participants) | 117 | 260
  Cognitive Functioning: Change at C3D1 | 0.9 (17.9) | -2.9 (19.1)
  Cognitive Functioning: Change at C4D1: number analyzed (Participants) | 100 | 231
  Cognitive Functioning: Change at C4D1 | 1.8 (18.9) | -1.7 (18.4)
  Cognitive Functioning: Change at C5D1: number analyzed (Participants) | 76 | 207
  Cognitive Functioning: Change at C5D1 | -1.5 (17.7) | -3.2 (17.7)
  Cognitive Functioning: Change at C6D1: number analyzed (Participants) | 66 | 171
  Cognitive Functioning: Change at C6D1 | -0.5 (18.5) | -2.8 (17.6)
  Cognitive Functioning: Change at C7D1: number analyzed (Participants) | 58 | 145
  Cognitive Functioning: Change at C7D1 | -2.3 (18.1) | -0.8 (18.8)
  Constipation: Baseline: number analyzed (Participants) | 160 | 312
  Constipation: Baseline | 15.8 (23.9) | 14.5 (23.7)
  Constipation: Change at C2D1: number analyzed (Participants) | 147 | 291
  Constipation: Change at C2D1 | 0.0 (24.0) | -6.0 (21.1)
  Constipation: Change at C3D1: number analyzed (Participants) | 117 | 260
  Constipation: Change at C3D1 | -2.3 (25.0) | -4.9 (20.8)
  Constipation: Change at C4D1: number analyzed (Participants) | 99 | 231
  Constipation: Change at C4D1 | -2.7 (24.6) | -5.5 (22.0)
  Constipation: Change at C5D1: number analyzed (Participants) | 76 | 207
  Constipation: Change at C5D1 | -1.3 (22.7) | -4.0 (21.0)
  Constipation: Change at C6D1: number analyzed (Participants) | 66 | 170
  Constipation: Change at C6D1 | -3.0 (27.3) | -3.5 (21.8)
  Constipation: Change at C7D1: number analyzed (Participants) | 58 | 145
  Constipation: Change at C7D1 | -4.6 (24.5) | -6.9 (22.5)
  Diarrhoea: Baseline: number analyzed (Participants) | 159 | 311
  Diarrhoea: Baseline | 6.3 (15.1) | 5.0 (14.4)
  Diarrhoea: Change at C2D1: number analyzed (Participants) | 147 | 292
  Diarrhoea: Change at C2D1 | -0.5 (17.9) | 10.2 (22.4)
  Diarrhoea: Change at C3D1: number analyzed (Participants) | 117 | 260
  Diarrhoea: Change at C3D1 | -0.9 (16.6) | 13.7 (26.3)
  Diarrhoea: Change at C4D1: number analyzed (Participants) | 100 | 231
  Diarrhoea: Change at C4D1 | -2.7 (21.0) | 13.1 (28.9)
  Diarrhoea: Change at C5D1: number analyzed (Participants) | 76 | 207
  Diarrhoea: Change at C5D1 | -2.6 (19.4) | 11.1 (27.7)
  Diarrhoea: Change at C6D1: number analyzed (Participants) | 66 | 171
  Diarrhoea: Change at C6D1 | -2.0 (17.4) | 14.0 (29.1)
  Diarrhoea: Change at C7D1: number analyzed (Participants) | 58 | 145
  Diarrhoea: Change at C7D1 | 1.1 (20.7) | 15.6 (30.9)
  Dyspnoea: Baseline: number analyzed (Participants) | 160 | 311
  Dyspnoea: Baseline | 15.0 (23.0) | 15.4 (22.2)
  Dyspnoea: Change at C2D1: number analyzed (Participants) | 146 | 291
  Dyspnoea: Change at C2D1 | 4.1 (23.5) | -2.1 (19.5)
  Dyspnoea: Change at C3D1: number analyzed (Participants) | 117 | 260
  Dyspnoea: Change at C3D1 | 2.8 (20.3) | 0.0 (20.9)
  Dyspnoea: Change at C4D1: number analyzed (Participants) | 100 | 231
  Dyspnoea: Change at C4D1 | 0.7 (23.2) | 0.0 (23.3)
  Dyspnoea: Change at C5D1: number analyzed (Participants) | 76 | 207
  Dyspnoea: Change at C5D1 | 2.6 (26.5) | 1.6 (23.2)
  Dyspnoea: Change at C6D1: number analyzed (Participants) | 66 | 170
  Dyspnoea: Change at C6D1 | 3.0 (26.6) | 0.2 (23.4)
  Dyspnoea: Change at C7D1: number analyzed (Participants) | 58 | 145
  Dyspnoea: Change at C7D1 | 1.7 (24.5) | -2.1 (21.2)
  Emotional Functioning: Baseline: number analyzed (Participants) | 160 | 312
  Emotional Functioning: Baseline | 73.1 (22.1) | 71.9 (22.1)
  Emotional Functioning: Change at C2D1: number analyzed (Participants) | 147 | 292
  Emotional Functioning: Change at C2D1 | 4.0 (17.9) | 5.1 (18.5)
  Emotional Functioning: Change at C3D1: number analyzed (Participants) | 117 | 260
  Emotional Functioning: Change at C3D1 | 4.5 (19.1) | 2.3 (21.6)
  Emotional Functioning: Change at C4D1: number analyzed (Participants) | 100 | 231
  Emotional Functioning: Change at C4D1 | 4.5 (18.5) | 2.6 (19.7)
  Emotional Functioning: Change at C5D1: number analyzed (Participants) | 76 | 207
  Emotional Functioning: Change at C5D1 | 5.2 (20.1) | -0.4 (21.8)
  Emotional Functioning: Change at C6D1: number analyzed (Participants) | 66 | 171
  Emotional Functioning: Change at C6D1 | 2.1 (20.5) | 2.4 (21.6)
  Emotional Functioning: Change at C7D1: number analyzed (Participants) | 58 | 145
  Emotional Functioning: Change at C7D1 | 5.3 (20.7) | 2.8 (19.7)
  Fatigue: Baseline: number analyzed (Participants) | 160 | 312
  Fatigue: Baseline | 30.8 (22.5) | 30.8 (22.0)
  Fatigue: Change at C2D1: number analyzed (Participants) | 147 | 292
  Fatigue: Change at C2D1 | 2.0 (19.2) | -0.5 (18.8)
  Fatigue: Change at C3D1: number analyzed (Participants) | 117 | 260
  Fatigue: Change at C3D1 | -1.5 (19.5) | 1.8 (21.5)
  Fatigue: Change at C4D1: number analyzed (Participants) | 100 | 231
  Fatigue: Change at C4D1 | -0.2 (19.1) | 2.4 (21.9)
  Fatigue: Change at C5D1: number analyzed (Participants) | 76 | 207
  Fatigue: Change at C5D1 | -0.1 (20.8) | 2.8 (20.4)
  Fatigue: Change at C6D1: number analyzed (Participants) | 66 | 171
  Fatigue: Change at C6D1 | 3.3 (20.0) | 2.4 (20.5)
  Fatigue: Change at C7D1: number analyzed (Participants) | 58 | 145
  Fatigue: Change at C7D1 | 1.0 (20.0) | 1.8 (20.5)
  Financial Difficulties: Baseline: number analyzed (Participants) | 160 | 310
  Financial Difficulties: Baseline | 18.5 (25.8) | 19.2 (27.1)
  Financial Difficulties: Change at C2D1: number analyzed (Participants) | 147 | 287
  Financial Difficulties: Change at C2D1 | -1.1 (20.4) | -2.8 (21.4)
  Financial Difficulties: Change at C3D1: number analyzed (Participants) | 117 | 258
  Financial Difficulties: Change at C3D1 | -0.9 (24.9) | -1.6 (24.4)
  Financial Difficulties: Change at C4D1: number analyzed (Participants) | 100 | 230
  Financial Difficulties: Change at C4D1 | 0.7 (25.1) | -0.3 (23.7)
  Financial Difficulties: Change at C5D1: number analyzed (Participants) | 76 | 205
  Financial Difficulties: Change at C5D1 | -0.4 (28.0) | 0.3 (24.9)
  Financial Difficulties: Change at C6D1: number analyzed (Participants) | 66 | 169
  Financial Difficulties: Change at C6D1 | 5.6 (30.1) | 0.4 (23.6)
  Financial Difficulties: Change at C7D1: number analyzed (Participants) | 58 | 143
  Financial Difficulties: Change at C7D1 | -0.6 (26.1) | 2.1 (23.1)
  Global Health Status/ QoL: Baseline: number analyzed (Participants) | 160 | 311
  Global Health Status/ QoL: Baseline | 65.2 (18.4) | 67.4 (20.3)
  Global Health Status/ QoL: Change at C2D1: number analyzed (Participants) | 147 | 291
  Global Health Status/ QoL: Change at C2D1 | -0.1 (16.7) | 1.0 (19.9)
  Global Health Status/ QoL: Change at C3D1: number analyzed (Participants) | 117 | 259
  Global Health Status/ QoL: Change at C3D1 | -1.0 (18.5) | -1.5 (20.9)
  Global Health Status/ QoL: Change at C4D1: number analyzed (Participants) | 100 | 230
  Global Health Status/ QoL: Change at C4D1 | -1.5 (18.6) | -1.6 (20.3)
  Global Health Status/ QoL: Change at C5D1: number analyzed (Participants) | 76 | 207
  Global Health Status/ QoL: Change at C5D1 | 0.3 (19.9) | -2.8 (20.3)
  Global Health Status/ QoL: Change at C6D1: number analyzed (Participants) | 66 | 171
  Global Health Status/ QoL: Change at C6D1 | -1.6 (18.6) | -3.4 (19.5)
  Global Health Status/ QoL: Change at C7D1: number analyzed (Participants) | 58 | 145
  Global Health Status/ QoL: Change at C7D1 | -1.1 (18.9) | -1.0 (18.9)
  Insomnia: Baseline: number analyzed (Participants) | 160 | 311
  Insomnia: Baseline | 26.0 (27.6) | 26.5 (27.7)
  Insomnia: Change at C2D1: number analyzed (Participants) | 146 | 289
  Insomnia: Change at C2D1 | -0.9 (24.4) | -3.8 (23.7)
  Insomnia: Change at C3D1: number analyzed (Participants) | 117 | 260
  Insomnia: Change at C3D1 | -3.4 (30.1) | -4.1 (26.4)
  Insomnia: Change at C4D1: number analyzed (Participants) | 100 | 231
  Insomnia: Change at C4D1 | -4.0 (28.9) | -1.0 (26.8)
  Insomnia: Change at C5D1: number analyzed (Participants) | 76 | 206
  Insomnia: Change at C5D1 | -0.4 (29.1) | -3.9 (25.6)
  Insomnia: Change at C6D1: number analyzed (Participants) | 66 | 170
  Insomnia: Change at C6D1 | -2.0 (30.3) | -2.4 (28.2)
  Insomnia: Change at C7D1: number analyzed (Participants) | 57 | 145
  Insomnia: Change at C7D1 | -4.1 (28.2) | -1.8 (27.2)
  Nausea/Vomiting: Baseline: number analyzed (Participants) | 160 | 312
  Nausea/Vomiting: Baseline | 5.9 (13.4) | 6.7 (13.7)
  Nausea/Vomiting: Change at C2D1: number analyzed (Participants) | 147 | 292
  Nausea/Vomiting: Change at C2D1 | 0.1 (11.9) | 1.6 (18.1)
  Nausea/Vomiting: Change at C3D1: number analyzed (Participants) | 117 | 260
  Nausea/Vomiting: Change at C3D1 | 0.7 (15.2) | 2.2 (17.6)
  Nausea/Vomiting: Change at C4D1: number analyzed (Participants) | 100 | 231
  Nausea/Vomiting: Change at C4D1 | 0.3 (17.9) | 2.3 (18.6)
  Nausea/Vomiting: Change at C5D1: number analyzed (Participants) | 76 | 207
  Nausea/Vomiting: Change at C5D1 | -1.1 (18.3) | 0.5 (15.4)
  Nausea/Vomiting: Change at C6D1: number analyzed (Participants) | 66 | 171
  Nausea/Vomiting: Change at C6D1 | 1.5 (18.0) | -0.6 (15.9)
  Nausea/Vomiting: Change at C7D1: number analyzed (Participants) | 58 | 145
  Nausea/Vomiting: Change at C7D1 | 2.6 (15.5) | 2.2 (18.8)
  Pain: Baseline: number analyzed (Participants) | 160 | 312
  Pain: Baseline | 28.0 (25.4) | 27.1 (24.9)
  Pain: Change at C2D1: number analyzed (Participants) | 147 | 292
  Pain: Change at C2D1 | -0.2 (24.0) | -5.0 (20.8)
  Pain: Change at C3D1: number analyzed (Participants) | 117 | 260
  Pain: Change at C3D1 | -3.7 (23.3) | -3.5 (22.6)
  Pain: Change at C4D1: number analyzed (Participants) | 100 | 231
  Pain: Change at C4D1 | -3.2 (24.7) | -1.7 (24.2)
  Pain: Change at C5D1: number analyzed (Participants) | 76 | 207
  Pain: Change at C5D1 | -3.3 (24.2) | -4.3 (22.9)
  Pain: Change at C6D1: number analyzed (Participants) | 66 | 171
  Pain: Change at C6D1 | -1.0 (23.0) | -2.2 (22.5)
  Pain: Change at C7D1: number analyzed (Participants) | 58 | 145
  Pain: Change at C7D1 | 0.3 (23.5) | -4.4 (19.8)
  Physical Functioning: Baseline: number analyzed (Participants) | 160 | 311
  Physical Functioning: Baseline | 76.7 (19.9) | 78.4 (18.8)
  Physical Functioning: Change at C2D1: number analyzed (Participants) | 147 | 292
  Physical Functioning: Change at C2D1 | -1.1 (13.4) | 1.6 (12.7)
  Physical Functioning: Change at C3D1: number analyzed (Participants) | 117 | 260
  Physical Functioning: Change at C3D1 | 2.0 (14.1) | 0.8 (15.7)
  Physical Functioning: Change at C4D1: number analyzed (Participants) | 100 | 231
  Physical Functioning: Change at C4D1 | 1.5 (16.1) | 0.3 (15.7)
  Physical Functioning: Change at C5D1: number analyzed (Participants) | 76 | 207
  Physical Functioning: Change at C5D1 | 2.0 (17.7) | 1.0 (13.5)
  Physical Functioning: Change at C6D1: number analyzed (Participants) | 66 | 171
  Physical Functioning: Change at C6D1 | 0.9 (18.4) | 1.1 (14.9)
  Physical Functioning: Change at C7D1: number analyzed (Participants) | 58 | 145
  Physical Functioning: Change at C7D1 | 1.6 (16.2) | 0.6 (14.2)
  Role Functioning: Baseline: number analyzed (Participants) | 160 | 312
  Role Functioning: Baseline | 79.1 (24.6) | 78.7 (24.0)
  Role Functioning: Change at C2D1: number analyzed (Participants) | 147 | 292
  Role Functioning: Change at C2D1 | -2.0 (19.3) | 1.7 (21.5)
  Role Functioning: Change at C3D1: number analyzed (Participants) | 117 | 260
  Role Functioning: Change at C3D1 | -0.4 (23.4) | -1.0 (23.9)
  Role Functioning: Change at C4D1: number analyzed (Participants) | 100 | 231
  Role Functioning: Change at C4D1 | 0.3 (23.0) | 0.4 (24.2)
  Role Functioning: Change at C5D1: number analyzed (Participants) | 76 | 207
  Role Functioning: Change at C5D1 | 1.8 (22.5) | -1.6 (21.6)
  Role Functioning: Change at C6D1: number analyzed (Participants) | 66 | 171
  Role Functioning: Change at C6D1 | -1.3 (23.8) | -1.6 (23.4)
  Role Functioning: Change at C7D1: number analyzed (Participants) | 58 | 145
  Role Functioning: Change at C7D1 | -0.3 (22.6) | 0.0 (22.9)
  Social Functioning: Baseline: number analyzed (Participants) | 160 | 312
  Social Functioning: Baseline | 83.2 (21.8) | 81.2 (23.1)
  Social Functioning: Change at C2D1: number analyzed (Participants) | 147 | 292
  Social Functioning: Change at C2D1 | -0.8 (19.9) | 2.7 (20.0)
  Social Functioning: Change at C3D1: number analyzed (Participants) | 117 | 259
  Social Functioning: Change at C3D1 | 1.3 (21.9) | -0.8 (23.2)
  Social Functioning: Change at C4D1: number analyzed (Participants) | 100 | 231
  Social Functioning: Change at C4D1 | 1.8 (18.2) | -0.5 (21.3)
  Social Functioning: Change at C5D1: number analyzed (Participants) | 76 | 207
  Social Functioning: Change at C5D1 | 0.9 (19.4) | -1.0 (23.3)
  Social Functioning: Change at C6D1: number analyzed (Participants) | 66 | 170
  Social Functioning: Change at C6D1 | -0.8 (20.1) | -1.6 (23.4)
  Social Functioning: Change at C7D1: number analyzed (Participants) | 58 | 145
  Social Functioning: Change at C7D1 | 0.6 (21.2) | 0.1 (19.7)

18. Secondary Outcome: Change From Baseline in Modified EORTC Quality of Life Questionnaire Breast Cancer Module 23 (QLQ-BR23) Score
Description: EORTC-QLQ-BR23 is a 23-item breast cancer-specific companion module to the EORTC-QLQ-C30 and consists of functional scales (body image, sexual enjoyment, sexual functioning, future perspective [FP]) and symptom scales (systemic side effects [SE], upset by hair loss, arm symptoms, breast symptoms). Questions used a 4-point scale (1=not at all, 2=a little, 3=quite a bit, 4=very much). Scores were averaged and transformed to a 0-100 scale. Higher scores for the functional scales indicated a higher/better level of functioning/healthy functioning. Higher scores for the symptom scales indicated worse symptoms.
Time Frame: Baseline, C2D1 up to C7D1 (each cycle=28 days)
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo+Fulvestrant | Taselisib+Fulvestrant
Number analyzed (Participants) | 176 | 340
score on a scale
  Arm Symptoms: Baseline: number analyzed (Participants) | 152 | 304
  Arm Symptoms: Baseline | 15.5 (18.8) | 19.3 (21.1)
  Arm Symptoms: Change at C2D1: number analyzed (Participants) | 140 | 282
  Arm Symptoms: Change at C2D1 | 0.1 (17.4) | -5.4 (15.6)
  Arm Symptoms: Change at C3D1: number analyzed (Participants) | 111 | 250
  Arm Symptoms: Change at C3D1 | -0.7 (19.5) | -6.1 (17.4)
  Arm Symptoms: Change at C4D1: number analyzed (Participants) | 95 | 219
  Arm Symptoms: Change at C4D1 | -1.4 (21.9) | -5.8 (15.8)
  Arm Symptoms: Change at C5D1: number analyzed (Participants) | 72 | 203
  Arm Symptoms: Change at C5D1 | 0.8 (17.0) | -6.6 (15.7)
  Arm Symptoms: Change at C6D1: number analyzed (Participants) | 63 | 167
  Arm Symptoms: Change at C6D1 | 1.1 (20.8) | -5.0 (18.5)
  Arm Symptoms: Change at C7D1: number analyzed (Participants) | 57 | 140
  Arm Symptoms: Change at C7D1 | -1.2 (19.7) | -6.0 (15.2)
  Body Image: Baseline: number analyzed (Participants) | 149 | 300
  Body Image: Baseline | 82.0 (21.7) | 80.8 (22.5)
  Body Image: Change at C2D1: number analyzed (Participants) | 135 | 276
  Body Image: Change at C2D1 | 1.8 (14.9) | 1.5 (16.5)
  Body Image: Change at C3D1: number analyzed (Participants) | 106 | 242
  Body Image: Change at C3D1 | 1.6 (18.0) | 1.1 (20.6)
  Body Image: Change at C4D1: number analyzed (Participants) | 92 | 214
  Body Image: Change at C4D1 | 1.1 (17.8) | 1.8 (20.6)
  Body Image: Change at C5D1: number analyzed (Participants) | 68 | 198
  Body Image: Change at C5D1 | 0.2 (19.5) | 0.0 (17.5)
  Body Image: Change at C6D1: number analyzed (Participants) | 60 | 164
  Body Image: Change at C6D1 | 1.1 (21.0) | 0.4 (18.2)
  Body Image: Change at C7D1: number analyzed (Participants) | 54 | 137
  Body Image: Change at C7D1 | 5.6 (18.8) | -0.3 (18.2)
  Breast Symptoms: Baseline: number analyzed (Participants) | 151 | 304
  Breast Symptoms: Baseline | 8.7 (14.6) | 11.0 (14.1)
  Breast Symptoms: Change at C2D1: number analyzed (Participants) | 139 | 282
  Breast Symptoms: Change at C2D1 | 0.0 (13.7) | -3.0 (11.8)
  Breast Symptoms: Change at C3D1: number analyzed (Participants) | 112 | 250
  Breast Symptoms: Change at C3D1 | -0.8 (13.3) | -3.5 (11.6)
  Breast Symptoms: Change at C4D1: number analyzed (Participants) | 95 | 220
  Breast Symptoms: Change at C4D1 | 0.1 (14.2) | -3.0 (11.8)
  Breast Symptoms: Change at C5D1: number analyzed (Participants) | 72 | 203
  Breast Symptoms: Change at C5D1 | -0.9 (14.5) | -2.0 (11.7)
  Breast Symptoms: Change at C6D1: number analyzed (Participants) | 63 | 167
  Breast Symptoms: Change at C6D1 | 1.7 (16.0) | -2.0 (12.9)
  Breast Symptoms: Change at C7D1: number analyzed (Participants) | 57 | 140
  Breast Symptoms: Change at C7D1 | 0.3 (12.6) | -3.2 (13.1)
  Future Perspective: Baseline: number analyzed (Participants) | 152 | 303
  Future Perspective: Baseline | 47.4 (31.5) | 47.3 (29.6)
  Future Perspective: Change at C2D1: number analyzed (Participants) | 139 | 281
  Future Perspective: Change at C2D1 | 3.4 (30.1) | 6.8 (27.4)
  Future Perspective: Change at C3D1: number analyzed (Participants) | 111 | 247
  Future Perspective: Change at C3D1 | 5.1 (29.5) | 4.3 (30.5)
  Future Perspective: Change at C4D1: number analyzed (Participants) | 95 | 220
  Future Perspective: Change at C4D1 | 6.0 (30.7) | 7.0 (29.2)
  Future Perspective: Change at C5D1: number analyzed (Participants) | 72 | 202
  Future Perspective: Change at C5D1 | 6.0 (30.3) | 5.0 (26.8)
  Future Perspective: Change at C6D1: number analyzed (Participants) | 63 | 167
  Future Perspective: Change at C6D1 | 6.9 (28.8) | 9.0 (31.4)
  Future Perspective: Change at C7D1: number analyzed (Participants) | 57 | 139
  Future Perspective: Change at C7D1 | 12.9 (29.4) | 7.0 (30.2)
  Sexual Enjoyment: Baseline: number analyzed (Participants) | 27 | 61
  Sexual Enjoyment: Baseline | 51.9 (26.7) | 62.8 (26.6)
  Sexual Enjoyment: Change at C2D1: number analyzed (Participants) | 17 | 35
  Sexual Enjoyment: Change at C2D1 | 5.9 (21.2) | 0.0 (18.1)
  Sexual Enjoyment: Change at C3D1: number analyzed (Participants) | 14 | 26
  Sexual Enjoyment: Change at C3D1 | 4.8 (22.1) | 1.3 (24.0)
  Sexual Enjoyment: Change at C4D1: number analyzed (Participants) | 8 | 24
  Sexual Enjoyment: Change at C4D1 | -8.3 (15.4) | 4.2 (24.7)
  Sexual Enjoyment: Change at C5D1: number analyzed (Participants) | 7 | 26
  Sexual Enjoyment: Change at C5D1 | -4.8 (23.0) | 2.6 (29.7)
  Sexual Enjoyment: Change at C6D1: number analyzed (Participants) | 5 | 17
  Sexual Enjoyment: Change at C6D1 | -6.7 (14.9) | -5.9 (24.3)
  Sexual Enjoyment: Change at C7D1: number analyzed (Participants) | 5 | 14
  Sexual Enjoyment: Change at C7D1 | -13.3 (29.8) | 9.5 (20.4)
  Sexual Functioning: Baseline: number analyzed (Participants) | 142 | 291
  Sexual Functioning: Baseline | 89.6 (17.9) | 89.9 (17.3)
  Sexual Functioning: Change at C2D1: number analyzed (Participants) | 126 | 267
  Sexual Functioning: Change at C2D1 | 1.6 (11.0) | 1.5 (14.2)
  Sexual Functioning: Change at C3D1: number analyzed (Participants) | 98 | 235
  Sexual Functioning: Change at C3D1 | 1.4 (10.6) | 1.8 (15.6)
  Sexual Functioning: Change at C4D1: number analyzed (Participants) | 86 | 203
  Sexual Functioning: Change at C4D1 | 1.9 (15.4) | 1.6 (13.9)
  Sexual Functioning: Change at C5D1: number analyzed (Participants) | 63 | 186
  Sexual Functioning: Change at C5D1 | -0.8 (20.6) | 2.6 (15.1)
  Sexual Functioning: Change at C6D1: number analyzed (Participants) | 55 | 156
  Sexual Functioning: Change at C6D1 | 2.4 (18.8) | 2.7 (15.0)
  Sexual Functioning: Change at C7D1: number analyzed (Participants) | 49 | 132
  Sexual Functioning: Change at C7D1 | 2.7 (18.1) | 2.3 (15.7)
  Systematic Therapy SEs: Baseline: number analyzed (Participants) | 152 | 304
  Systematic Therapy SEs: Baseline | 15.7 (14.2) | 14.7 (12.0)
  Systematic Therapy SEs: Change at C2D1: number analyzed (Participants) | 140 | 282
  Systematic Therapy SEs: Change at C2D1 | 0.2 (11.4) | 2.5 (11.0)
  Systematic Therapy SEs: Change at C3D1: number analyzed (Participants) | 112 | 250
  Systematic Therapy SEs: Change at C3D1 | 1.2 (14.4) | 4.0 (13.6)
  Systematic Therapy SEs: Change at C4D1: number analyzed (Participants) | 95 | 220
  Systematic Therapy SEs: Change at C4D1 | 1.5 (13.2) | 4.0 (13.3)
  Systematic Therapy SEs: Change at C5D1: number analyzed (Participants) | 72 | 203
  Systematic Therapy SEs: Change at C5D1 | 2.4 (13.8) | 5.5 (14.1)
  Systematic Therapy SEs: Change at C6D1: number analyzed (Participants) | 63 | 167
  Systematic Therapy SEs: Change at C6D1 | 2.9 (15.2) | 5.7 (15.6)
  Systematic Therapy SEs: Change at C7D1: number analyzed (Participants) | 57 | 140
  Systematic Therapy SEs: Change at C7D1 | 3.5 (16.7) | 4.8 (15.0)
  Upset by Hair Loss: Baseline: number analyzed (Participants) | 33 | 63
  Upset by Hair Loss: Baseline | 23.2 (28.2) | 27.0 (29.2)
  Upset by Hair Loss: Change at C2D1: number analyzed (Participants) | 14 | 31
  Upset by Hair Loss: Change at C2D1 | -11.9 (28.1) | -4.3 (22.3)
  Upset by Hair Loss: Change at C3D1: number analyzed (Participants) | 13 | 29
  Upset by Hair Loss: Change at C3D1 | -7.7 (30.9) | 0.0 (26.7)
  Upset by Hair Loss: Change at C4D1: number analyzed (Participants) | 13 | 27
  Upset by Hair Loss: Change at C4D1 | 2.6 (16.5) | 0.0 (29.2)
  Upset by Hair Loss: Change at C5D1: number analyzed (Participants) | 8 | 28
  Upset by Hair Loss: Change at C5D1 | 0.0 (25.2) | 10.7 (27.3)
  Upset by Hair Loss: Change at C6D1: number analyzed (Participants) | 6 | 26
  Upset by Hair Loss: Change at C6D1 | 11.1 (27.2) | 16.7 (30.2)
  Upset by Hair Loss: Change at C7D1: number analyzed (Participants) | 8 | 26
  Upset by Hair Loss: Change at C7D1 | 4.2 (11.8) | 14.1 (32.9)

ADVERSE EVENTS:
Time Frame: From randomization up to the end of study, approximately 6.2 years
Description: All-cause mortality was reported based on the ITT population: all randomized participants regardless of whether they received any amount of study treatment. Serious and non-serious adverse events were reported based on the safety-evaluable population: all randomized participants who received at least one dose of taselisib, placebo or fulvestrant regardless of the PIK3CA-mutation status of their tumors with participants allocated to the treatment arm associated with the regimen actually received.
Arm/Group | Placebo+Fulvestrant | Taselisib+Fulvestrant
All-Cause Mortality (participants affected / at risk) | 100/214 | 197/417
Serious Adverse Events (participants affected / at risk) | 23/213 | 154/416
Other Adverse Events (participants affected / at risk) | 183/213 | 396/416
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo+Fulvestrant (N=213) | Taselisib+Fulvestrant (N=416)
ANAEMIA (Blood and lymphatic system disorders) | 1 (2) | 2 (2)
PANCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0) | 2 (2)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 0 (0) | 1 (1)
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 1 (1)
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 (0) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 1 (1)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 (0) | 1 (1)
ALCOHOLIC PANCREATITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
COLITIS (Gastrointestinal disorders) | 0 (0) | 16 (17)
DIARRHOEA (Gastrointestinal disorders) | 0 (0) | 37 (40)
DYSPEPSIA (Gastrointestinal disorders) | 0 (0) | 1 (1)
DYSPHAGIA (Gastrointestinal disorders) | 0 (0) | 1 (1)
ENTERITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
ENTEROCOLITIS (Gastrointestinal disorders) | 0 (0) | 3 (3)
GASTRIC ULCER (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTRITIS (Gastrointestinal disorders) | 0 (0) | 2 (2)
NAUSEA (Gastrointestinal disorders) | 2 (2) | 4 (5)
OESOPHAGEAL ULCER (Gastrointestinal disorders) | 0 (0) | 1 (1)
OESOPHAGITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
PANCREATITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
PANCREATITIS ACUTE (Gastrointestinal disorders) | 0 (0) | 2 (2)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 2 (3)
STOMATITIS (Gastrointestinal disorders) | 0 (0) | 2 (2)
VOMITING (Gastrointestinal disorders) | 1 (1) | 4 (4)
ASTHENIA (General disorders) | 0 (0) | 1 (1)
CHEST DISCOMFORT (General disorders) | 0 (0) | 2 (2)
CHEST PAIN (General disorders) | 0 (0) | 3 (3)
CHILLS (General disorders) | 1 (1) | 0 (0)
DEATH (General disorders) | 1 (1) | 3 (3)
FATIGUE (General disorders) | 1 (1) | 2 (2)
MUCOSAL INFLAMMATION (General disorders) | 0 (0) | 1 (1)
PAIN (General disorders) | 1 (1) | 0 (0)
PYREXIA (General disorders) | 2 (2) | 3 (3)
SWELLING FACE (General disorders) | 1 (1) | 0 (0)
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 0 (0) | 1 (1)
CHOLELITHIASIS (Hepatobiliary disorders) | 0 (0) | 1 (1)
HEPATOTOXICITY (Hepatobiliary disorders) | 0 (0) | 1 (1)
ANAPHYLACTIC SHOCK (Immune system disorders) | 0 (0) | 1 (1)
APPENDICITIS PERFORATED (Infections and infestations) | 0 (0) | 1 (1)
ATYPICAL MYCOBACTERIAL PNEUMONIA (Infections and infestations) | 0 (0) | 1 (1)
BRONCHITIS (Infections and infestations) | 0 (0) | 1 (1)
CELLULITIS (Infections and infestations) | 0 (0) | 2 (2)
CHOLERA (Infections and infestations) | 0 (0) | 1 (1)
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 0 (0) | 1 (1)
CYSTITIS ESCHERICHIA (Infections and infestations) | 0 (0) | 1 (1)
DIARRHOEA INFECTIOUS (Infections and infestations) | 0 (0) | 3 (3)
ENTEROCOLITIS INFECTIOUS (Infections and infestations) | 0 (0) | 2 (2)
GASTROENTERITIS (Infections and infestations) | 0 (0) | 1 (1)
GASTROENTERITIS VIRAL (Infections and infestations) | 0 (0) | 1 (1)
HERPES ZOSTER (Infections and infestations) | 0 (0) | 1 (1)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1)
PNEUMONIA (Infections and infestations) | 1 (1) | 10 (10)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1)
SEPSIS (Infections and infestations) | 1 (1) | 5 (5)
SEPTIC ARTHRITIS STAPHYLOCOCCAL (Infections and infestations) | 0 (0) | 1 (2)
SKIN INFECTION (Infections and infestations) | 0 (0) | 2 (2)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 3 (3)
UROSEPSIS (Infections and infestations) | 0 (0) | 1 (1)
VIRAL INFECTION (Infections and infestations) | 0 (0) | 1 (1)
CLAVICLE FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
FALL (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
HIP FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
JOINT DISLOCATION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
TOXICITY TO VARIOUS AGENTS (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
WRIST FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1) | 2 (2)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1) | 1 (1)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 1 (1) | 0 (0)
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
DEHYDRATION (Metabolism and nutrition disorders) | 1 (1) | 7 (7)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 7 (7)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
COCCYDYNIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OSTEONECROSIS OF JAW (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
RHABDOMYOLYSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
HEPATOCELLULAR CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
INTRACRANIAL TUMOUR HAEMORRHAGE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
CEREBRAL HAEMATOMA (Nervous system disorders) | 0 (0) | 1 (1)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 2 (2) | 1 (1)
FACIAL PARALYSIS (Nervous system disorders) | 1 (1) | 0 (0)
HEADACHE (Nervous system disorders) | 0 (0) | 3 (3)
HYPOAESTHESIA (Nervous system disorders) | 0 (0) | 2 (2)
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 0 (0) | 1 (1)
TRIGEMINAL NEURALGIA (Nervous system disorders) | 0 (0) | 1 (1)
VITH NERVE PARALYSIS (Nervous system disorders) | 1 (1) | 0 (0)
CONFUSIONAL STATE (Psychiatric disorders) | 0 (0) | 1 (1)
MENTAL STATUS CHANGES (Psychiatric disorders) | 0 (0) | 2 (2)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0 (0) | 4 (4)
HAEMATURIA (Renal and urinary disorders) | 0 (0) | 1 (1)
RENAL FAILURE (Renal and urinary disorders) | 0 (0) | 1 (1)
URETEROLITHIASIS (Renal and urinary disorders) | 1 (1) | 0 (0)
INTERMENSTRUAL BLEEDING (Reproductive system and breast disorders) | 0 (0) | 1 (1)
ACUTE RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (2)
PLEURITIC PAIN (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 10 (10)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
DRUG ERUPTION (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
PRURITUS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
RASH (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
TOXIC SKIN ERUPTION (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
EMBOLISM (Vascular disorders) | 0 (0) | 1 (1)
EMBOLISM VENOUS (Vascular disorders) | 0 (0) | 1 (1)
HYPERTENSION (Vascular disorders) | 0 (0) | 1 (1)
SHOCK (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo+Fulvestrant (N=213) | Taselisib+Fulvestrant (N=416)
ANAEMIA (Blood and lymphatic system disorders) | 20 (23) | 44 (62)
NEUTROPENIA (Blood and lymphatic system disorders) | 9 (12) | 28 (39)
ABDOMINAL PAIN (Gastrointestinal disorders) | 20 (25) | 55 (67)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 8 (8) | 31 (35)
CONSTIPATION (Gastrointestinal disorders) | 32 (36) | 32 (36)
DIARRHOEA (Gastrointestinal disorders) | 45 (76) | 255 (602)
DRY MOUTH (Gastrointestinal disorders) | 18 (19) | 55 (62)
DYSPEPSIA (Gastrointestinal disorders) | 5 (5) | 32 (51)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 4 (4) | 23 (25)
NAUSEA (Gastrointestinal disorders) | 54 (71) | 154 (233)
STOMATITIS (Gastrointestinal disorders) | 8 (11) | 87 (139)
VOMITING (Gastrointestinal disorders) | 25 (41) | 86 (116)
ASTHENIA (General disorders) | 40 (65) | 77 (104)
FATIGUE (General disorders) | 40 (51) | 105 (134)
MUCOSAL INFLAMMATION (General disorders) | 11 (15) | 44 (67)
OEDEMA PERIPHERAL (General disorders) | 11 (13) | 19 (25)
PYREXIA (General disorders) | 9 (10) | 48 (61)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 11 (17) | 33 (41)
URINARY TRACT INFECTION (Infections and infestations) | 9 (10) | 38 (50)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 9 (13) | 36 (47)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 15 (19) | 35 (47)
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 12 (12) | 15 (17)
BLOOD CREATININE INCREASED (Investigations) | 6 (7) | 25 (28)
WEIGHT DECREASED (Investigations) | 6 (6) | 42 (50)
DECREASED APPETITE (Metabolism and nutrition disorders) | 23 (25) | 119 (136)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 21 (26) | 166 (233)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 2 (2) | 31 (37)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 35 (50) | 69 (95)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 28 (32) | 62 (82)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 17 (19) | 24 (26)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 6 (8) | 32 (34)
MYALGIA (Musculoskeletal and connective tissue disorders) | 14 (14) | 36 (42)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 19 (27) | 33 (42)
DIZZINESS (Nervous system disorders) | 18 (23) | 46 (58)
DYSGEUSIA (Nervous system disorders) | 5 (5) | 36 (41)
HEADACHE (Nervous system disorders) | 27 (38) | 88 (122)
INSOMNIA (Psychiatric disorders) | 18 (19) | 37 (40)
COUGH (Respiratory, thoracic and mediastinal disorders) | 34 (41) | 64 (78)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 17 (17) | 50 (53)
ALOPECIA (Skin and subcutaneous tissue disorders) | 6 (6) | 50 (53)
DRY SKIN (Skin and subcutaneous tissue disorders) | 10 (10) | 37 (40)
PRURITUS (Skin and subcutaneous tissue disorders) | 18 (28) | 52 (75)
RASH (Skin and subcutaneous tissue disorders) | 17 (24) | 80 (116)
HOT FLUSH (Vascular disorders) | 27 (27) | 24 (26)
HYPERTENSION (Vascular disorders) | 11 (16) | 33 (42)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-24): https://cdn.clinicaltrials.gov/large-docs/21/NCT02340221/Prot_SAP_000.pdf